CLINICAL TRIAL: NCT02912910
Title: Changes in Central Arterial Pressure When Comparing Nifedipine and Labetalol for Routine Hypertension Control in Pregnancy
Brief Title: Changes in Central Arterial Pressure When Comparing Nifedipine/Labetalol for Routine Hypertension Control in Pregnancy
Status: Withdrawn | Type: Observational
Why Stopped: PI withdrew protocol
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Jennifer Goldkamp, MD, MD, St. Louis University
Other Study IDs: 27464
Record Dates: First submitted 2016-09-12; First posted 2016-09-23 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nifedipine; Labetalol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Nifedipine: patients will be assigned to antihypertensive medications by their physicians in the course of their routine care
  Interventions: Other: Nifedipine
- Labetalol: patients will be assigned to antihypertensive medications by their physicians in the course of their routine care
  Interventions: Other: Labetalol

INTERVENTIONS:
Other: Nifedipine — patients will be assigned to antihypertensive medications by their physicians in the course of their routine care
  Groups: Nifedipine
Other: Labetalol — patients will be assigned to antihypertensive medications by their physicians in the course of their routine care
  Groups: Labetalol

SUMMARY:
To study central blood pressure changes caused by commonly used high blood pressure medications in pregnancy.

DETAILED DESCRIPTION:
Central blood pressures in addition to pulse wave velocity will be attained prior to medication, and then every 30 minutes for 4 hours (total of 9 readings). Sphygmomanometer readings will be completed at the same time (total readings 9). These readings are all related to the study.

Nursing will have the opportunity to to record the routine sphygmomanometer readings for their routine vitals if they chose to do so.

Their participation will be complete after the 4 hour assessment is complete.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Women with hypertensive disease in pregnancy who are currently being treated with nifedipine xl or labetalol

Exclusion Criteria:

* Multiple pregnancy
* Currently on multiple anti-hypertension medications
* Narcotic use
* Irregular heart rhythms or arrhythmias
* Peripheral arterial disease, leg artery disease
* Reynaud's phenomena
* Intense cold/hypothermia
* If there is a wound at location of where central arterial cuff would be placed or tonometer for carotid assessment
* Known sensitivity to labetalol or nifedipine
* Severe tachycardia (>120)
* Greater than 1st degree heart block
* Severe asthma
* Congestive heart failure or heart disease
* Lupus
* Inability to adequately monitor BP
* Currently receiving magnesium sulfate

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women in our clinics in addition to admitted to our antepartum units will be screened for inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-09 (Estimated); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
central blood pressure changes | every 30 min for 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Goldkamp, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No